CLINICAL TRIAL: NCT06871527
Title: Fruquintinib Combined With Tislelizumab and FOLFOX as First-Line Treatment For Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma: A Single-center, Open-label, Phase Ib/II Clinical Study
Brief Title: Fruquintinib Combined With PD-1 Inhibitor and FOLFOX as First-Line Treatment For Advanced Gastric Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025ZSLYEC-081
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Gastric (Stomach) Cancer; Gastric Adenocarcinoma; Fruquintinib; PD-1 Inhibitor; Tislelizumab; GEJ Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — HMPL-013; tislelizumab; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fruquintinib + tislelizumab + FOLFOX (Experimental): fruquintinib + tislelizumab + FOLFOX
  Interventions: Drug: fruquintinib + tislelizumab + FOLFOX

INTERVENTIONS:
Drug: fruquintinib + tislelizumab + FOLFOX — phase Ib: fruquintinib (3+3 dose escalation design): L1: 3 mg/d, L2: 4 mg/d, L3: 5 mg/d, qd po, D1-14, Q3W; tislelizumab: 200mg, I.V., D1, Q2W; 5-Fluorouracil: 400mg/m2, D1, followed by 2400 mg/m2 as a continuous IV infusion over 46 hours,Q2W; leucovorin : 400mg/m2, I.V., D1, Q2W; Oxaliplatin: 85mg/m2, ivgtt 2h, D1, Q2W.
  phase II: fruquintinib: RP2D; tislelizumab: 200mg, I.V., D1, Q2W; 5-Fluorouracil: 400mg/m2, D1, followed by 2400 mg/m2 as a continuous IV infusion over 46 hours,Q2W; leucovorin: 400mg/m2, I.V., D1, Q2W; Oxaliplatin: 85mg/m2, ivgtt 2h, D1, Q2W.

SUMMARY:
This study was designed to explore the efficacy and safety of fruquintinib combined with tislelizumab and FOLFOX regimen as the first treatment (first-line) for adults diagnosed with locally advanced unresectable or metastatic gastric or gastroesophageal junction (GEJ) adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old (including 18 and 75 years old);
* Eastern Cooperation Oncology Group (ECOG) performance status of 0-1;
* Pathologically determined gastric or gastroesophageal junction adenocarcinoma;
* Advanced patients with radiographic confirmation of inoperable complete resection;
* No previous anti-tumor treatment for metastatic diseases;
* At least one measurable lesion according to RECIST version 1.1;
* Ability to take medications orally;
* No active bleeding;
* Adequate organ functions:

Absolute neutrophil count ≥2×109/L; Platelet ≥100×109/L; Hemoglobin ≥90g/L; WBC≥4×109/L Total bilirubin ≤ 1.5XULN; ALT and AST ≤2.5XULN ； Serum creatinine (Cr) ≤1.5XULN；

• Have fully understood the study and voluntarily signed the informed consent;

Exclusion Criteria:

* Patients who had received any drug in the study protocol in the last year;
* Deficient mismatch repair (dMMR) or MSI-H detected by genetic test;
* HER2 positive（HER-2 3+, or HER-2 2+ and FISH+）;
* Hypertension that could not be controlled by drugs before enrollment was defined as: systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥90 mmHg;
* Patients with acute coronary syndromes (including myocardial infarction and unstable angina) received coronary angioplasty or stenting within 6 months before enrollment;
* Patients with massive pleural or peritoneal effusion requiring drainage;
* Patients with severe ECG abnormalities or heart diseases (such as cardiac insufficiency, myocardial infarction, angina pectoris) that affect clinical treatment;
* Severe lung diseases (such as interstitial pneumonia, pulmonary fibrosis, severe emphysema, etc.);
* Mental disorders or central nervous system diseases or brain metastases affecting clinical treatment;
* Patients with autoimmune diseases;
* Patients with grade 3 or higher bleeding within 4 weeks;
* Patients with a history of allergy to any drug, similar drug or vehicle in this study;
* Had a major surgical procedure (thoracotomy, or laparotomy , etc.) within 4 weeks prior to the first dose of study therapy;
* Patients with nonhealed wounds, ulcers, or fractures;
* Patients who required systemic corticosteroids (excluding temporary testing, prophylactic administration for anaphylaxis), or immunosuppressive agents or had received such agents within 14 days before enrollment;
* Pregnant or lactating women, or patients of childbearing age who refused contraception during the study period;
* Investigators believe that the patient has any other conditions that are not suitable for participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Maximum tolerated dose (MTD) | At the end of Cycle 1 (each cycle is 21 days)
  Maximum Tolerated Dose (MTD) of fruquintinib. Investigators leading the study will find the maximum tolerated dose by assessing the rate of serious side effects (known as "dose limiting toxicities") among participants according to the CTCAE 5.0.
Phase Ib: RD | At the end of Cycle 1 (each cycle is 21 days)
  To determine the recommended phase 2 dose of fruquintinib, according to the dose limiting toxicities (DLTs).
Six-month progression-free survival | At six months
  The proportion of patients who remain alive and free from disease progression for at least 6 months after initiating treatment.

SECONDARY OUTCOMES:
PFS | Up to 3 years
  PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first.
OS | Up to 3 years
  OS is defined as the time from the date of randomization to the date of death due to any cause.
ORR | Up to 3 years
  ORR is defined as the percentage of patients with a best overall response of complete response (CR) or partial response (PR) per RESISTv1.1.
DCR | Up to 3 years
  DCR is defined as the percentage of patients with a best overall response of confirmed complete or partial response, or stable disease (CR+ PR + SD) per RESISTv1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided